CLINICAL TRIAL: NCT05771272
Title: Investigation of the Relationship Between Low Back and Back Line of the Lower Extremity Flexibility and Rowing Performance on Elite Rowers
Brief Title: The Relationship Between Flexibility and Rowing Performance on Elite Rowers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: TCİl
Record Dates: First submitted 2023-02-14; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Flexibility; Performance
Keywords: Rowing Performance; Low back flexibility; Hamstring flexibility; Ankle flexibility; Rowing
MeSH Terms: interventions — Sitting Position

STUDY DESIGN:
Intervention Model Description: All rower sport player were assessed by CAIT , lower extremity flexibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elite Rowers (Other): They are young men rowers aged between 16-18 years, rowing age of at least 2 years, and continuing to row sport actively.
  Interventions: Diagnostic Test: Sit and Reach Test; Diagnostic Test: Weight Bearing Lunge Test

INTERVENTIONS:
Diagnostic Test: Sit and Reach Test — To conduct the test, a box measuring 32 centimeters in height, 45 centimeters in width, and 35 cm in length, and the upper surface of the box was 15 cm longer than the area on which the feet rest. The participant is positioned on the ground with both legs fully extended, separated by shoulder width, and flat on the box. The participant positioned themselves with one hand on top of the other, knees fully extended, stretched as far forward as they could, sliding their hands across the ruler's top, and kept that posture for at least two seconds. The end location of the fingertips on or approaching the ruler was measured in centimeters to get the sit and reach score. Scores that are higher showed improved performance. The best result is recorded after the test was run three times.
Diagnostic Test: Weight Bearing Lunge Test — To conduct the test, with a tape measure on the floor, measure the distance from the big toe's end to the wall. Participants make a lunging motion forward until their knee hit on the wall. The participant's foot is positioned on the floor with the big toe and heel line aligned on the tape measure. To determine how close to the wall a subject could touch the wall with their knee while still keeping their heel in contact. The tape measure is then used to calculate the distance from the big toe's tip to the wall in centimeters. Increasing the distance indicates that the participant has less ankle dorsiflexion range
  Other Names: Dorsiflexion Lunge Test

SUMMARY:
The aim of the research is to examine the effects of ankle, low back and hamstring flexibility of young male rowers on 2000-m rowing performance. Research data were collected on January 8, 2023, at Turkey Indoor Rowing Championship. The subjects of the research (n=26) is young male rowers aged 16-18 and with at least 2 years of rowing age. Outcome measures in this study are 'Sit and Reach Test' and 'Weight Bearing Lunge Test'.

DETAILED DESCRIPTION:
The aim of the research is to examine the effects of ankle, low back and hamstring flexibility of young male rowers on 2000-m rowing performance. Research data were collected on January 8, 2023, at Turkey Indoor Rowing Championship.The study included 26 male rowers who competed in different Turkish rowing teams. The subjects completed a form requesting certain personal and training data also consent form was filled. After subject completed the form, flexibility of the back and backline of lower extremities were measured. To measure the low back and hamstring muscle flexibility, 'sit and reach test' and assess the ankle flexibility 'weight bearing lunge test' were conducted on each rower. In order to measure performance of rowers, the time results of 2000-m ergometer test were recorded after the race.

ELIGIBILITY:
Inclusion Criteria:

* Continuing to rowing sport actively
* Rowing age of at least 2 years
* Young men rowers aged between the 16-18 years

Exclusion Criteria:

* Acute injury in the lumbar region and lower extremity and/or presence of pain for more than 3 months,
* Surgical operation in the lumbar region and lower extremity region in the last 6 months,
* Over 18 years old or under 16 years old and less than 2 years of rowing age

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2023-01-08 (Actual)

PRIMARY OUTCOMES:
Sit and Reach Test | 1 day
  The Sit and Reach Test is one of the linear flexibility tests that helps determine how extensible the hamstrings and lower back are. In a study, the test was used to measure flexibility of rowers. The box measured 32 centimeters in height, 45 centimeters in width, and 35 cm in length and the upper surface of box was 15 cm longer than the area on which the feet rest. The subject was positioned on the ground with both legs fully extended, separated by shoulder-width, and flat on the box. The participant positioned themselves with one hand on top of the other, knees fully extended, stretched as far forward as they could, sliding their hands across the ruler's top, and kept that posture for at least two seconds. The end location of the fingertips on or approaching the ruler was measured in centimeters to get the sit and reach score. Scores that were higher showed improved performance. The best result recorded after the test was run three times.
Weight Bearing Lunge Test | 1 day
  The Weight-Bearing Lunge Test, also known as the Dorsiflexion Lunge Test, is used to measure the ankle joint's dorsiflexion range of motion. With a tape measure on the floor, measure the distance from the big toe's end to the wall. Subjects made a lunging motion forward until their knee hit on the wall. The subject's foot was positioned on the floor with the big toe and heel line aligned on the tape measure. To determine how close to the wall a subject could touch the wall with their knee while still keeping their heel in contact. The tape measure was then used to calculate the distance from the big toe's tip to the wall in centimeter. Increasing the distance indicates that the subject has less ankle dorsi flexion range

CONTACTS AND LOCATIONS:
Overall Officials: Elif T Çil, PhD, Study Director — Yeditepe University; Can Seçinti, BSc, Principal Investigator — Yeditepe University; Çağatay Şekeröz, Principal Investigator — Yeditepe University; Yağmur Barlas, BSc, Principal Investigator — Yeditepe University; Deniz Özlüer, BSc, Principal Investigator — Yeditepe University
Locations (1):
- Turkish Rowing Federation, Istanbul, Kadıköy, Turkey (Türkiye)